CLINICAL TRIAL: NCT01574144
Title: Observational Study of Reducing 30-day Admissions in Post-discharge Subjects
Brief Title: REducing 30-day ADMIssions in posT-discharge Subjects (READMIT)
Acronym: READMIT-HF
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: READMIT-HF
Record Dates: First submitted 2012-04-03; First posted 2012-04-10 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AVIVO™ PiiX Patch Monitor System: Heart failure patients monitored continuously for 30 days post-discharge.
  Interventions: Device: AVIVO™ PiiX Patch Monitor System

INTERVENTIONS:
Device: AVIVO™ PiiX Patch Monitor System — External monitoring for 30 days post-discharge.

SUMMARY:
The purpose of this observational study is to collect and characterize multiple physiologic data from a broad subset of subjects with acute heart failure (HF)

Changes in physiologic data are expected to correlate with 30-day readmission rates in this population

DETAILED DESCRIPTION:
This is a multi-center, non-randomized feasibility study aimed at obtaining data from systolic and diastolic HF subjects in the hospital, with continued monitoring using an external wearable monitor for up to 4 weeks post-hospital-discharge. Data will be collected during the hospital stay and at in office follow-up visits at 1 week and 1 month post-hospital discharge

The data will help generate hypotheses and aid in determining whether development of a detection algorithm for acute heart failure decompensation is feasible. Due to the feasibility nature of this study there is no minimum required sample size but it is anticipated that the study will enroll up to 100 subjects from seven (7) study sites in the United States and one (1) study site in Australia

The study objectives are:

* Collect and characterize physiologic data from subjects with acute decompensated heart failure.
* Characterization of data related to health care utilizations within 30-days Post-discharge
* Correlation between patch monitor collected data and inpatient clinical data
* Correlation between patch monitor data and other clinical data collected after patient discharge (30-60 days)

ELIGIBILITY:
Inclusion Criteria:

* Subject with acute decompensated heart failure
* Subject (or legal guardian) willing to give consent for their participation
* Subject ≥18 years of age

Exclusion Criteria:

* Subject who is expected to receive a heart transplant or a ventricular assist device within 6 months
* Subject who cannot tolerate placement of external patch monitor on chest in the proposed location (ECG Lead II orientation)
* Subject with known allergies or hypersensitivities to adhesives or hydrogels
* Subject with implantable devices with active minute ventilation sensors.
* Subject who will not comply to study protocol requirements. This includes completing required data collection, and attending required follow up study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients who are admitted to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: READMIT-HF Study Team, Study Director — Medtronic
Locations (8):
- United States (7):
  - Scripps Green Hospital, La Jolla, California
  - Bay Area Cardiology, Tampa, Florida
  - United Heart and Cardiovascular, Saint Paul, Minnesota
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Mohawk Valley Heart Institute, Utica, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee
- The Alfred Hospital, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVIVO™ PiiX Patch Monitor System
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrollment
Arm/Group | AVIVO™ PiiX Patch Monitor System
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 60
  Australia | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Health Care Utilizations
Description: Percentage of Participants with health care utilizations. Healthcare utilizations include hospitalizations, urgent care visits and emergency department visits.
Time Frame: 30 days post-discharge
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AVIVO™ PiiX Patch Monitor System
Number analyzed (Participants) | 70
percentage of participants | 28.6 [18.4 to 40.6]

2. Secondary Outcome: Change in Body Weight Per Unit Change in Thoracic Impedance
Description: Change in body weight per unit change in thoracic impedance. The regression coefficients between body weight and thoracic impedance.
Time Frame: Discharge to 30 days post discharge
Population: All subjects with changes of body weight and impedance from discharge to 30 days post discharge.
Measure: Mean (95% Confidence Interval); unit: lbs/Ohm
Groups:
- Heart Failure Patients Monitored Continuously With AVIVO PiiX: AVIVO™ PiiX Patch Monitor System: External monitoring from enrollment to discharge: regression coefficient
Arm/Group | Heart Failure Patients Monitored Continuously With AVIVO PiiX
Number analyzed (Participants) | 54
lbs/Ohm | -0.03 [-0.15 to 0.09]

ADVERSE EVENTS:
Time Frame: From enrollment to 3 months post-discharge
Description: An adverse event (AE) is considered a serious AE if it
  1. Lead to death OR
  2. Lead to a serious deterioration in subject's health (life threatening illness/injury, permanent impairment of body, hospitalization/prolonged, medical/surgical intervention to prevent the previously mentioned conditions) OR
  3. Lead to fetal distress/death/defect
Arm/Group | AVIVO™ PiiX Patch Monitor System
Serious Adverse Events (participants affected / at risk) | 14/70
Other Adverse Events (participants affected / at risk) | 9/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVIVO™ PiiX Patch Monitor System (N=70)
Atrial Fribrillation (Cardiac disorders) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 1 (1)
Cardiac Failure congrestive (Cardiac disorders) | 4 (4)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
HyperKalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Mental Status Changes (Psychiatric disorders) | 2 (2)
Renal Failure Chronic (Renal and urinary disorders) | 1 (1)
Scrotal Oedema (Reproductive system and breast disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVIVO™ PiiX Patch Monitor System (N=70)
Cardiac Failure congestive (Cardiac disorders) | 3 (3)
Application Site Bruise (General disorders) | 1 (1)
Application Site Rash (General disorders) | 2 (2)
Blood Thyroid Stimlating Hormone Increased (Investigations) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No